CLINICAL TRIAL: NCT06567860
Title: Characterizing Late-season Influenza Vaccine Responses to Compare the 2023 and 2024 Vaccine Formulations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: La Jolla Institute for Immunology (Other)
Responsible Party: Principal Investigator, Tal Einav, Assistant Professor, La Jolla Institute for Immunology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 286
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Influenza A
Keywords: Influenza vaccine; Immune response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Late season influenza vaccine (Experimental): Every participant receives the 2023 influenza vaccine between May-June 2024, and then the 2024 influenza vaccine in September-October 2024. Blood draws are taken at Day 0, 30, and 90 post-vaccination.
  Interventions: Biological: Influenza Fluzone vaccine

INTERVENTIONS:
Biological: Influenza Fluzone vaccine — Fluzone vaccine administered in both May-June and in September-October for each participant.

SUMMARY:
Every 1-2 years, the seasonal influenza vaccine composition changes to include updated viruses, yet the precise effects of updating the vaccine remain understudied. Since the vaccine formulation for each season (with a season defined as starting in July and ending the following June) expires on June 30, vaccine formulations cannot be compared head-to-head. Thus, the 2023 and 2024 vaccines have only been compared by analyzing people given the former vaccine in the fall of 2023 and people given the latter vaccine in the fall of 2024, and baseline repertoires may have greatly changed over the course of that year. To that end, the investigators will vaccinate a cohort with the 2023 influenza vaccine between May-June 2024, in order to compare responses between individuals receiving the 2023 vaccine last fall, the 2023 vaccine late in the season (this cohort), and the 2024 vaccine next fall. The investigators will further assess whether the late-season 2023 vaccine primed this cohort to respond better to the standard 2024 vaccine with standard timing (vaccine administered around September-October).

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-64 years of age
* Males or non-pregnant, non-nursing females
* Weigh at least 85 pounds for whole blood draw
* Ability to provide signed informed consent
* Subjects must plan to receive the intramuscular influenza vaccine at the La Jolla Institute for Immunology

Exclusion Criteria:

* Received an influenza vaccine in the past year
* Infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
* History of certain anemias
* Presence of significant cardiovascular disease, systemic diseases including, but not limited to, diabetes which is not controlled, renal disease, liver disease, malignancy, infection, or blood clotting disorder
* Inability to provide informed consent
* Recent whole blood donation within 56 days or leukapheresis within 112 days
* Children (under 18 years of age), elderly (65 years of age or older), pregnant or nursing females
* Individuals with egg allergies
* Has ever had Guillain-Barré syndrome

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Einav, PhD, Principal Investigator — La Jolla Institute for Immunology
Locations (1):
- La Jolla Institute for Immunology, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be included in all relevant publications.
Supporting Information: Analytic Code
Time Frame: Data will be available upon publication.
Access Criteria: Data will be available with no restrictions.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were recruited into either Arm 1 (receiving only the late-season 2023 vaccine) or Arm 2 (receiving the late-season 2023 vaccine and then the 2024 vaccine three months later). 9 participants chose to participate in Arm 1 and 14 in Arm 2.
Groups:
- Arm 1: Late-season 2023 Influenza Vaccine: Participants that had not been previously vaccinated for influenza during the 2023-24 season (i.e. no influenza vaccine since July 1, 2023) were given the 2023 vaccine in either May or June of 2024. Antibody HAI responses were measured 0, 30, and 90 days following this vaccination.
- Arm 2: Late-season 2023 Influenza Vaccine Followed by the 2024 Influenza Vaccine: As in Arm 1, participants that had not been previously vaccinated for influenza during the 2023-24 season were given the 2023 vaccine in either May or June of 2024. Antibody HAI responses were measured 0, 30, and 90 days following this vaccination. Following that, participants were given the 2024 influenza vaccine in September, October, or November of 2024. Antibody HAI responses were measured 0, 30, and 90 days following this vaccination.
Period: Overall Study
Arm/Group | Arm 1: Late-season 2023 Influenza Vaccine | Arm 2: Late-season 2023 Influenza Vaccine Followed by the 2024 Influenza Vaccine
Started | 9 | 14
Completed | 9 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Late-season 2023 Influenza Vaccine | Arm 2: Late-season 2023 Influenza Vaccine Followed by the 2024 Influenza Vaccine | Total
Number analyzed (Participants) | 9 | 14 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30 (9) | 28 (5) | 29 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 3 | 10 | 13
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Antibody Response After the Late-season 2023 Vaccine
Description: The antibody response will be measured by hemagglutination inhibition (HAI) in adults between 18 and 64 years old who have not had an influenza vaccination prior to the study.
Time Frame: 0, 30, and 90 days after the 2023 vaccine
Population: HAI titers were computed for all participants in each arm at every time point using the geometric mean and the geometric standard deviation, E^(standard deviation of log(titers)). For example, the value of 6±1.4 for Arm 1's H1N1 day 0 measurement should be interpreted as a geometric mean of 6, and a 1.4x standard error (so that values were generally between 6/1.4 and 6×1.4).
Measure: Geometric Mean (Standard Deviation); unit: HAI Titer
Arm/Group | Arm 1: Late-season 2023 Influenza Vaccine | Arm 2: Late-season 2023 Influenza Vaccine Followed by the 2024 Influenza Vaccine
Number analyzed (Participants) | 9 | 14
HAI Titer
  H1N1, Day 0 | 6 (1.4) | 6 (1.5)
  H1N1, Day 30 | 74 (4.8) | 27 (4.1)
  H1N1, Day 90 | 40 (5.1) | 21 (3.8)
  H3N2, Day 0 | 10 (2.8) | 9 (2.1)
  H3N2, Day 30 | 43 (5.2) | 42 (3.2)
  H3N2, Day 90 | 34 (5.4) | 28 (2.6)
  B Victoria, Day 0 | 8 (1.6) | 10 (1.9)
  B Victoria, Day 30 | 54 (2.5) | 57 (2.6)
  B Victoria, Day 90 | 34 (2.1) | 46 (2.7)
  B Yamagata, Day 0 | 47 (5.2) | 46 (4.0)
  B Yamagata, Day 30 | 254 (2.8) | 145 (3.2)
  B Yamagata, Day 90 | 148 (3.4) | 88 (3.0)

2. Primary Outcome: Magnitude of the Antibody Response After the 2024 Vaccine
Description: The antibody response will be measured by hemagglutination inhibition (HAI) in adults between 18 and 64 years old who have not had an influenza vaccination prior to the study. This outcome was only performed on Arm 2.
Time Frame: Day 0, 30, and 90 after the 2024 vaccine
Population: Serum was only collected for Arm 2 participants.
Measure: Geometric Mean (Standard Error); unit: HAI Titer
Arm/Group | Arm 1: Late-season 2023 Influenza Vaccine | Arm 2: Late-season 2023 Influenza Vaccine Followed by the 2024 Influenza Vaccine
Number analyzed (Participants) | 0 | 14
HAI Titer
  H1N1, Day 0 |  | 16 (3.7)
  H1N1, Day 30 |  | 18 (3.6)
  H1N1, Day 90 |  | 16 (3.5)
  H3N2, Day 0 |  | 21 (3.0)
  H3N2, Day 30 |  | 31 (2.6)
  H3N2, Day 90 |  | 26 (2.8)
  B Victoria, Day 0 |  | 31 (2.7)
  B Victoria, Day 30 |  | 76 (2.3)
  B Victoria, Day 90 |  | 47 (2.1)
  B Yamagata, Day 0 |  | 80 (3.2)
  B Yamagata, Day 30 |  | 84 (3.6)
  B Yamagata, Day 90 |  | 55 (3.2)

ADVERSE EVENTS:
Time Frame: From receipt of the 2023 vaccine (day 0) through study completion, an average of 3 months for Arm 1 and 7 months for Arm 2.
Arm/Group | Arm 1: Late-season 2023 Influenza Vaccine | Arm 2: Late-season 2023 Influenza Vaccine Followed by the 2024 Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT06567860/Prot_000.pdf
  • Informed Consent Form (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT06567860/ICF_001.pdf